CLINICAL TRIAL: NCT00286208
Title: A Randomized Study of Sublingual Versus Oral Misoprostol Administration Following Mifepristone 200 mg for Abortion up to 63 Days Gestation
Brief Title: Study of Sublingual Versus Oral Misoprostol Administration Following Mifepristone 200 mg for Abortion up to 63 Days Gestation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.1.5
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Induced Abortion
Keywords: Medical abortion; mifepristone; misoprostol
MeSH Terms: interventions — Mifepristone; Misoprostol

ARMS (2):
- Sublingual Misoprostol (Active Comparator): 400 mcg of sublingual misoprostol
  Interventions: Drug: Mifepristone, misoprostol
- Oral Misoprostol (Active Comparator): Misoprostol administered orally
  Interventions: Drug: Mifepristone, misoprostol

INTERVENTIONS:
Drug: Mifepristone, misoprostol

SUMMARY:
This open-label, randomized study is being conducted to determine whether a dose of 400 mcg of sublingual misoprostol (i.e., under the tongue) taken 24 hours following administration of mifepristone 200 mg is effective and acceptable at inducing an abortion compared with misoprostol taken orally.

The goal of this study is to provide answers to the following four questions:

1. Is a regimen of medical abortion with mifepristone using sublingual misoprostol at least as effective as using oral misoprostol up to 63 days since the last menstrual period (LMP)?
2. Are the side effects with sublingual use tolerable for women?
3. Is sublingual administration of misoprostol acceptable to women?
4. Is one of the regimens (sublingual or oral) superior in terms of efficacy, safety (side-effects) or acceptability?

ELIGIBILITY:
Inclusion Criteria:

* Women presenting for medical abortion who consent to participate
* Possibility of final gestational age of less than or equal to 63 days
* General good health
* Willing to provide contact information for purposes of follow-up

Exclusion Criteria:

* Conditions which contraindicate the use of mifepristone or misoprostol
* Women presenting for medical abortion who do not consent to participate

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1443 (Actual)
Dates: Start 2005-08; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Need for surgical completion for incomplete abortions or ongoing viable pregnancies at follow up visit Study day 15. | 2 weeks after mifepristone administration

SECONDARY OUTCOMES:
Side effects | 48 hours
Acceptability for women | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Raghavan, M.Sc., Study Director — Gynuity Health Projects; Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects; Rasha Dabash, MPH, Study Director — Gynuity Health Projects; Selma Hajri, MD, Principal Investigator — Reproductive Health Consultant; Ayse Akin, MD, MPH, Principal Investigator — Baskent University; Ilana Dzuba, MHS, Study Director — Gynuity Health Projects
Locations (9):
- State University of Medicine and Pharmacy, Chisinau, Moldova
- Tunisia (4):
  - Centre de Planification Familiale de l'Ariana, Aryanah
  - Centre de Planification Familiale la Bardo, Tunis
  - Maternité de La Rabta, Tunis
  - Private clinic, Tunis
- Turkey (Türkiye) (4):
  - Dr. Zekai Tahir Burak Women's Health Training and Research Hospital, Ankara
  - MoH Ankara Etlik Maternity and Gyneacological Training Hospital, Ankara
  - Haydarpaşa Numune Training and Research Hospital Family Planning Clinic, Istanbul
  - Ege Maternity and Gyneacological Training and Research Hospital, Izmir